CLINICAL TRIAL: NCT04106193
Title: Addressing Intimate Partner Violence Among Women Veterans: Evaluating the Impact and Effectiveness of VHA's Response
Brief Title: Addressing Intimate Partner Violence Among Women Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: SDR 18-150; Iverson Miller SDR (Other: VA Boston Healthcare System)
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Intimate Partner Violence
Keywords: intimate partner violence; women Veterans; screening; primary care

STUDY DESIGN:
Intervention Model Description: Hybrid type II implementation-effectiveness design; stepped wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toolkit + Implementation as Usual (Experimental): Participating clinics assigned to this arm will receive a guiding toolkit and implementation as usual regarding IPV screening practices.
  Interventions: Other: Implementation as usual; Other: Toolkit
- Toolkit + Blended Facilitation (Experimental): Participating clinics assigned to this arm will receive a guiding toolkit and blended facilitation to support IPV screening practices.
  Interventions: Other: Blended Facilitation; Other: Toolkit

INTERVENTIONS:
Other: Blended Facilitation — Blended facilitation consists of an External Facilitator and Internal Facilitator to support adoption of intimate partner violence screening practices for WVs treated in primary care.
  Arms: Toolkit + Blended Facilitation
Other: Implementation as usual — Implementation as usual refers to traditional, site-initiated support for screening practices to detect intimate partner violence among WVs treated in primary care.
  Arms: Toolkit + Implementation as Usual
Other: Toolkit — All study arms will feature a toolkit meant to guide sites' adoption of intimate partner violence screening among WVs treated in primary care.

SUMMARY:
Up to 20% of women Veterans (WV) using VHA primary care experience past-year intimate partner violence (IPV), which contributes to numerous physical and mental health conditions, including suicidality. Despite national recommendations to screen WVs for IPV, there is low adoption of IPV screening programs in primary care. In response, VHA is spreading IPV screening programs in Women's Health Model 1 and Model 2 primary care clinics, where the majority of WV VHA primary care patients receive care. The systematic and effective implementation of IPV screening programs within primary care clinics is expected to enhance care for WVs as well as improve access to, and timeliness of, IPV-related care. Given the high prevalence of IPV among WVs and its significant negative health effects, successful implementation of IPV screening programs is expected to reduce morbidity among WV VHA patients. This stepped wedge hybrid II implementation/effectiveness study will assess efforts to implement routine IPV screening for WV VHA patients.

DETAILED DESCRIPTION:
Background: Intimate partner violence (IPV) is common among women Veterans (WVs), with nearly 20% of WVs treated in Veterans Health Administration (VHA) primary care clinics experiencing past-year IPV. VHA's Women's Health Services (WHS), the IPV Assistance Program, and the Offices of Primary Care and Mental Health and Suicide Prevention developed recommendations for implementing IPV screening programs in primary care. More than two-thirds of WV primary care patients receive care in "Model 1" (i.e., mixed-gender primary care) and "Model 2" (i.e., separate but shared space) clinics, but uptake of screening is low in these clinics. WHS therefore plans to use Blended Facilitation (BF) to roll out IPV screening programs in Model 1 and Model 2 primary care clinics. Given the high number of these clinics throughout VHA, it is unclear whether resource-intensive BF is feasible and whether a less intensive strategy (i.e., toolkit + Implementation as Usual [IAU]) can be effective. Research is also needed on the clinical effectiveness of IPV screening programs.

Significance/Impact: Given the high prevalence of IPV among WVs and its significant health effects, successful implementation of IPV screening programs is expected to improve healthcare services and reduce morbidity among WV VHA patients, an HSR&D priority area.

Innovation: This study will be the most comprehensive evaluation of both the implementation impact and clinical effectiveness of IPV screening programs globally. It is innovative in its inclusion of four strong VHA operations partners dedicated to successful implementation of IPV screening programs. This project capitalizes on a time-sensitive opportunity to advance IPV screening programs and implementation science.

Specific Aims: This objective of this proposal is to comprehensively evaluate two strategies for implementing IPV screening programs through achieving three specific aims.

1. Evaluate the degree of reach, adoption, implementation fidelity, and maintenance achieved using two implementation strategies for IPV screening programs.
2. Evaluate the clinical effectiveness of IPV screening programs, as evidenced by disclosure rates and post-screening psychosocial service use.
3. Identify multi-level barriers to and facilitators of IPV screening program implementation and sustainment.

Methodology: The investigators propose a cluster randomized, stepped wedge, Hybrid Type II program evaluation design to compare the impact of two implementation strategies (BF + toolkit vs. toolkit + IAU) and the clinical effectiveness of IPV screening programs. This study will use a mixed methods approach to collect quantitative (clinical records data) and qualitative (key informant interviews) implementation outcomes (Aims 1 and 3), as well as quantitative (clinical records data) clinical effectiveness outcomes (Aim 2). The investigators will supplement these data collection methods with surveys to assess implementation strategies survey to be completed pre-BF, post-BF, and in the maintenance phase. The integrated-Promoting Action on Research Implementation in Health Services (i-PARIHS) framework will guide the qualitative data collection and analysis. Summative data will be analyzed using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) Framework.

Next Steps/Implementation: This study's four VHA operations partners are eager to use the study results to inform future implementation strategies and clinical practices to spread IPV screening programs to all VHA primary care clinics and other clinical settings so that this vital intervention is accessible to all WV VHA patients.

ELIGIBILITY:
Inclusion Criteria:

* Women Veterans age 18+
* Presenting for care at participating VA-based primary care clinics.
* Due to be screened for intimate partner violence (IPV)

Exclusion Criteria:

* IPV screen completed in past year.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient population is limited to Women Veterans (WVs) eligible for screening for intimate partner violence (IPV) in primary care.
Enrollment: 7421 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Reach (primary implementation outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of WVs seen in Model 1 and 2 clinics during the last three months of each study phase who receive IPV screening
Change in Disclosure Rate (primary clinical effectiveness outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of eligible WVs who screen positive for IPV

SECONDARY OUTCOMES:
Change in Psychosocial Service Use (secondary clinical effectiveness outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of WVs accepting psychosocial service referrals following a positive IPV screen who use such services within two months
Adoption of Screening (secondary implementation outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of PC clinics completing IPV screening with eligible WVs during evaluation periods
Change in Adoption of Referrals / Resource Provision (secondary implementation outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of PC clinics delivering IPV screening program to eligible WVs during evaluation periods, including evidence of resource provision and referral offered for those with positive screens
Change in Implementation Fidelity (secondary implementation outcome) | For each site, the proportion calculated at baseline (months 1-3) will be compared to the proportion calculated for the latter half of the facilitation period (months 7-9).
  Change in proportion of clinics for whom WVs accept referrals attend psychosocial services within two months of positive screen
Maintenance (secondary implementation outcome) | For each site, the proportion calculated in the latter half of the facilitation phase (months 7-9) will be compared to the proportion calculated for the last three months of the maintenance phase (months 19-21)
  Change in proportion of WVs seen in Model 1 and 2 clinics during the last three months of the facilitation and maintenance phases who receive IPV screening

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M. Iverson, PhD MA BA, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (10):
- United States (10):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Gulf Coast Veterans Health Care System, Biloxi, MS, Biloxi, Mississippi
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - Jonathan M. Wainwright Memorial VA Medical Center, Walla Walla, WA, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iverson KM, Dichter ME, Stolzmann K, Adjognon OL, Lew RA, Bruce LE, Gerber MR, Portnoy GA, Miller CJ. Assessing the Veterans Health Administration's response to intimate partner violence among women: protocol for a randomized hybrid type 2 implementation-effectiveness trial. Implement Sci. 2020 May 7;15(1):29. doi: 10.1186/s13012-020-0969-0. PMID 32381013
- [Result] Ogden SN, Dichter ME, Bazzi AR. Intimate partner violence as a predictor of substance use outcomes among women: A systematic review. Addict Behav. 2022 Apr;127:107214. doi: 10.1016/j.addbeh.2021.107214. Epub 2021 Dec 18. PMID 34933089
- [Derived] Adjognon OL, Brady JE, Iverson KM, Stolzmann K, Dichter ME, Lew RA, Gerber MR, Portnoy GA, Iqbal S, Haskell SG, Bruce LAE, Miller CJ. Using the Matrixed Multiple Case Study approach to identify factors affecting the uptake of IPV screening programs following the use of implementation facilitation. Implement Sci Commun. 2023 Nov 21;4(1):145. doi: 10.1186/s43058-023-00528-x. PMID 37990345
- [Derived] Iverson KM, Stolzmann KL, Brady JE, Adjognon OL, Dichter ME, Lew RA, Gerber MR, Portnoy GA, Iqbal S, Haskell SG, Bruce LE, Miller CJ. Integrating Intimate Partner Violence Screening Programs in Primary Care: Results from a Hybrid-II Implementation-Effectiveness RCT. Am J Prev Med. 2023 Aug;65(2):251-260. doi: 10.1016/j.amepre.2023.02.013. Epub 2023 Apr 7. PMID 37031032